CLINICAL TRIAL: NCT05721404
Title: Icodextrin Postpones the Shift of Low Dose to Full Dose Dialysis in the First Year of Incremental Peritoneal Dialysis: A Randomized Controlled Trial
Brief Title: Icodextrin Postpones the Shift of Low Dose to Full Dose Dialysis in the First Year of Incremental Peritoneal Dialysis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Xiao Yang, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2022]042
Record Dates: First submitted 2023-02-04; First posted 2023-02-10 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Dialysis
Keywords: peritoneal dialysis; incremental peritoneal dialysis; icodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICO (icodextrin) (Experimental): When the extracellular water /total body water (ECW/TBW) ≥ 0.40, the patients in the ICO arm will be prescribed icodextrin (Extraneal) for long night dwell to improve fluid overload till their re-measurement of ECW/TBW < 0.40.
  Interventions: Drug: Icodextrin Peritoneal Dialysis Solution
- CON (control) (Other): When the extracellular water /total body water (ECW/TBW) ≥ 0.40, the patients in the CON arm will be prescribed hypertonic Dextrose solution for long night dwell to improve fluid overload till their ECW/TBW < 0.40
  Interventions: Drug: Hypertonic Dextrose solution

INTERVENTIONS:
Drug: Icodextrin Peritoneal Dialysis Solution — Icodextrin (Extraneal) for long night dwell
  Arms: ICO (icodextrin)
Drug: Hypertonic Dextrose solution — Hypertonic Dextrose solution for long night dwell
  Arms: CON (control)

SUMMARY:
We hypothesize incremental peritoneal dialysis (incremental PD) protocol with icodextrin solution will help patients to achieve adequate ultrafiltration and adequate dialysis with less glucose exposure by manipulating a low frequency of exchanges, therefore prolong the time from incremental protocol to full dose protocol (Full dose dialysis is defined as a dialysis dose of more than 8 L (4 exchanges of 2 L) per day). The goal of this clinical trial is to investigate the effect of icodextrin postponing the shift of low dose to full dose dialysis in the first year of incremental peritoneal dialysis. The main questions are:

* The effect of icodextrin on the shift of low dose to full dose dialysis in the first year in patients on incremental peritoneal dialysis.
* The effect of icodextrin on clinical outcomes in patients on incremental peritoneal dialysis, such as the first episode of peritonitis, the incidence of anuria, the first incidence of hospitalization, technical failure, all cause mortality, cardiovascular disease free survival and the quality of life.

Participants will be 1:1 randomized to the ICO (icodextrin) arm and CON (control) arm. Both arms patients will be followed every 2 months for fluid status by bioimpedance analysis. An extracellular water /total body water (ECW/TBW) ≥ 0.40 or edema is defined as overhydration (OH). The OH patients in the ICO arm will be prescribed icodextrin (Extraneal) for long night dwell to improve fluid overload till their re-measurement of ECW/TBW < 0.40 or edema disappeared. The OH patients in the CON arm will be prescribed hypertonic Dextrose solution for long night dwell to improve fluid overload till their ECW/TBW < 0.40 or edema disappeared.

Researchers will compare the time of transferring from low dose PD to full dose and the clinical outcomes in the first year between the patients in ICO and CON groups to see the effect of icodextrin on the shift of low dose to full dose dialysis and clinical outcomes in the first year in patients on incremental peritoneal dialysis. Successful completion of the study will advance our strategy of incremental PD and help to prolong the shift from incremental to full dose dialysis, and offer new opportunities for the development of an effective and economical therapy for PD patients with residual kidney function (RKF)

DETAILED DESCRIPTION:
Specific details of Treatment to be used in conducting study:

The objective of this study is to investigate the effects of icodextrin on postponing the shift of lowdose at the initial dialysis to full dose dialysis in the first year of PD in patients with incremental PD. The specific details of treatment/intervention are as follow:

1. Incident PD patients of SYSU PD center who meet the inclusion criteria will be recruited. All participants will be 1:1 randomized to the ICO (icodextrin) arm and CON (control) arm. Day 0 was defined as 6 weeks ± 4 weeks after CAPD initiation.
2. The patients in both the ICO and CON arms are prescribed Dextrose 2 L x 3 for incremental peritoneal dialysis during the first year.
3. Both arms patients will be followed every 2 months for fluid status by bioimpedance analysis (BIA). An extracellular water /total body water (ECW/TBW) ≥ 0.40 is defined as overhydration (OH).
4. The OH patients in the ICO arm will be prescribed icodextrin (Extraneal) for long night dwell to improve fluid overload till their re-measurement of ECW/TBW < 0.40 or edema disappeared. The OH patients in the CON arm will be prescribed hypertonic Dextrose solution for long night dwell to improve fluid overload till their ECW/TBW < 0.40 or edema disappeared. This means that all the patients in both arms will use the same three bags of glucose solution per day at the beginning of the study. When patients have overhydration [(ECW/TBW) ≥ 0.4 or edema], the long night dwell glucose solution in the ICO group will be replaced by Icodextrin till ECW/TBW < 0.40 or edema disappeared. While patients with overhydration in the CON group will increase glucose concentration till their ECW/TBW < 0.40 or edema disappeared. (The advantage of icodextrin has been proven in patients with ultrafiltration failure, high transport peritoneal membranes, and diabetics as compared to standard glucose based dialysate.
5. Both arms patients will be followed every 2 months for clinical manifestations, medication, and PD prescription (PD modality, dosage, and dialysate glucose concentration) during routine visits.
6. Patients in the both arms will be transferred to full dose dialysis if they have the following clinical manifestations: refractory fluid overload, unexplained nausea or vomiting, hyperkalemia, metabolic acidosis, uncontrollable hyperphosphatemia, uremia, neuropathy, pericarditis, sleep disorder, restless legs syndrome, pruritus, intractable anemia.
7. If necessary, medications will be used for treatment of hypertension, anaemia, chronic kidney disease-mineral and bone disorder, malnutrition, hyperlipidemia, the acid-base imbalance, electrolyte disturbance, etc.
8. If heart failure happened, patients in both the ICO and CON arms will be performed intermittent PD (IPD).

Efficacy Assessments:

1. Baseline data and follow-up information will be collected. Baseline demographics includes age, sex, primary kidney disease, body mass index (BMI), and diabetes. Baseline laboratory data include GFR, creatinine clearance (CrCl), urea clearance weekly (Kt/Vurea), ultrafiltration volume, systolic blood pressure (SBP), diastolic blood pressure (DBP), 24-h urine volume, serum albumin, serum creatinine (Scr), blood urea nitrogen (BUN), uric acid (UA), hemoglobin, intact parathyroid hormone (iPTH), total cholesterol, triglycerides, calcium, and phosphorus.
2. Both 24-hour urine and PD effluent will be collected at the same time each day to calculate Kt/Vurea, creatinine clearance, normalized protein clearance rate, and measured GFR using Adequest 2.0 software (Baxter Healthcare).
3. The adequacy of renal and peritoneal solute clearance will be assessed by total weekly Kt/V calculated using standard methodology. CAPD patients will receive Kt/V test every 2-4 months.
4. Peritoneal function and biomarkers for peritoneal biocompatibility will be performed: the peritoneal equilibration test (PET), sodium dip, CA125 and interleukin- 6 (IL-6) in effluent of patients in both groups.
5. All baseline data will be collected at day 0. Both arms patients will be followed up every 2 months for clinical manifestations, medication, and PD prescription (PD modality, dosage, and dialysate glucose concentration) during routine visits.
6. Events such as the episodes of peritonitis, transferring to hemodialysis (HD), anuria, cardiovascular disease(CVD), hospitalization, all cause death and CVD death will be recorded.
7. Quality of Life (Medical Outcomes Study 36-Item Short From Survey) will be measured and collected at the Day 0 and at the end of the study.

Statistical Methods:

1. Sample size:

   A preliminary analysis using database of our PD center showed: A total of 193 subjects (of which 97 are in group1 and 96 are in group 2) achieves 80% power at a 0.0500 significance level to detect a difference of 0.1900 between 0.6200 and 0.8100--the proportions surviving in groups 1 and 2, respectively. This corresponds to a hazard ratio of 0.4408. The proportion of patients lost during follow up was 0.0500. These results are based on the assumption that the hazard rates are proportional. Accordingly, 194 subjects (97 in each group) were intended to be included in the study.
2. Primary Endpoint Analysis:

   Primary endpoint (event that transferring from a low dose dialysis to full dose dialysis in the first year of incremental PD) analyses are on the basis of the intent-to-treat approach. Patient event-free survival will be calculated using the Kaplan-Meier method, and differences between different groups are assessed by log-rank tests. Considering patients transferred to other modalities as censoring (competing end points), the Fine and Gray proportional subhazards model will be used to create a competing risk model.
3. Secondary endpoint(s) analysis:

Secondary endpoints include first episode of peritonitis, anuria, CVD free survival, first hospitalization, technique failure (transferring to HD), all-cause and cardiovascular mortality, which will be evaluating using the Kaplan-Meier method, and differences between different groups are assessed by log-rank tests. Considering patients transferred to other modalities as censoring (competing end points), the Fine and Gray proportional subhazards model will be used to create a competing risk model. Quality of Life (PF, RP, BP, GH, VT, SF, RE, MH, PCS, MCS, total score of SF-36) will be evaluated using an unpaired Student's t test or Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* The estimated glomerular filtration rate (eGFR) ≥ 3ml/min·1.73m2 when enrolled;
* The 24-hour urine volume ≥ 500ml when enrolled;
* The patient or his lawful representative is able to receive and complete training of home peritoneal dialysis;
* Patients were able to follow the follow-up schedule and other requirements of the study;
* Patients can come to the peritoneal dialysis center for regular follow-up (once every 2 months or more);
* Participants were expected to remain on peritoneal dialysis for at least 13 months;
* Patients with good compliance;
* Informed consent was obtained.

Exclusion Criteria:

* Treated with both peritoneal dialysis and hemodialysis;
* Patients who have previously received a kidney transplant and have been receiving immunosuppressive therapy;
* Contraindications to bioelectrical impedance analysis (BIA) testing (e.g., amputation, use of a pacemaker or prosthesis);
* Allergy to Icodextrin, starch and starch products, or suffer from glycogen storage disease;
* Contraindications for the use of icodextrin;
* HIV-positive participants;
* Patients with tumors or other serious diseases have a life expectancy of less than one year;
* Mental illness that interferes with the patient's understanding of the test requirements and completion of the test process;
* Chronic wasting diseases such as tuberculosis, cirrhosis, hematological or other malignancies;
* Patients who are pregnant, intending to become pregnant, or breastfeeding during the study period;
* The patients had a history of drug abuse or alcoholism 2 years before the screening period;
* Patients who are unwilling or not expected to fully comply with the visits and evaluations required by the protocol;
* Patients who, in the investigator's judgment, have other serious or acute medical conditions that may prevent them from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The time that transferring from incremental PD to full dose in the first year of incremental PD | From date of randomization until the date of transferring from incremental PD to full dose, assessed up to 12 months
  The time of transferring to full dose dialysis was subtracted from the time of andomization

SECONDARY OUTCOMES:
The time of the first episode of peritonitis | From date of randomization until the date of first documented date of peritonitis, whichever came first, assessed up to 12 months
  The time of the first episode of peritonitis was subtracted from the time of randomization
The time of the incidence of anuria | From date of randomization until the date of first documented date of anuria, whichever came first, assessed up to 12 months
  The time of the incidence of anuria was subtracted from the time of randomization
The time of the first incidence of hospitalization | From date of randomization until the date of first documented date of hospitalization, whichever came first, assessed up to 12 months
  The time of the first incidence of hospitalization was subtracted from the time of randomization
The time of technical failure (transferring to HD) | From date of randomization until the date of first documented date of technical failure (transferring to HD), whichever came first, assessed up to 12 months
  The time of technical failure was subtracted from the time of randomization
All cause mortality and cardiovascular mortality | From date of randomization until the date of documented date of death due to cardiovascular cause and other causes, assessed up to 12 months
  The time of death was subtracted from the time of randomization
Cardiovascular disease free survival | From date of randomization until the date of first documented date of cardiovascular disease, whichever came first, assessed up to 12 months
  The time of the incidence of cardiovascular disease was subtracted from the time of randomization
The quality of life | Record patients' quality of life at the time of randomization and the first year after randomization
  Medical Outcomes Study 36-Item Short From Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Yang, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas B, Wulf S, Bikbov B, Perico N, Cortinovis M, Courville de Vaccaro K, Flaxman A, Peterson H, Delossantos A, Haring D, Mehrotra R, Himmelfarb J, Remuzzi G, Murray C, Naghavi M. Maintenance Dialysis throughout the World in Years 1990 and 2010. J Am Soc Nephrol. 2015 Nov;26(11):2621-33. doi: 10.1681/ASN.2014101017. Epub 2015 Jul 24. PMID 26209712
- [Background] Brown EA, Blake PG, Boudville N, Davies S, de Arteaga J, Dong J, Finkelstein F, Foo M, Hurst H, Johnson DW, Johnson M, Liew A, Moraes T, Perl J, Shroff R, Teitelbaum I, Wang AY, Warady B. International Society for Peritoneal Dialysis practice recommendations: Prescribing high-quality goal-directed peritoneal dialysis. Perit Dial Int. 2020 May;40(3):244-253. doi: 10.1177/0896860819895364. Epub 2020 Jan 21. No abstract available. PMID 32063219
- [Background] Lee Y, Chung SW, Park S, Ryu H, Lee H, Kim DK, Joo KW, Ahn C, Lee J, Oh KH. Incremental Peritoneal Dialysis May be Beneficial for Preserving Residual Renal Function Compared to Full-dose Peritoneal Dialysis. Sci Rep. 2019 Jul 12;9(1):10105. doi: 10.1038/s41598-019-46654-2. PMID 31300708
- [Background] Sandrini M, Vizzardi V, Valerio F, Ravera S, Manili L, Zubani R, Lucca BJ, Cancarini G. Incremental peritoneal dialysis: a 10 year single-centre experience. J Nephrol. 2016 Dec;29(6):871-879. doi: 10.1007/s40620-016-0344-z. Epub 2016 Aug 31. PMID 27582136
- [Background] Ankawi GA, Woodcock NI, Jain AK, Garg AX, Blake PG. The Use of Incremental Peritoneal Dialysis in a Large Contemporary Peritoneal Dialysis Program. Can J Kidney Health Dis. 2016 Dec 13;3:2054358116679131. doi: 10.1177/2054358116679131. eCollection 2016. PMID 28781885
- [Background] Yan H, Fang W, Lin A, Cao L, Ni Z, Qian J. Three Versus 4 Daily Exchanges and Residual Kidney Function Decline in Incident CAPD Patients: A Randomized Controlled Trial. Am J Kidney Dis. 2017 Apr;69(4):506-513. doi: 10.1053/j.ajkd.2016.08.019. Epub 2016 Oct 15. PMID 27751610
- [Background] Garofalo C, Borrelli S, De Stefano T, Provenzano M, Andreucci M, Cabiddu G, La Milia V, Vizzardi V, Sandrini M, Cancarini G, Cupisti A, Bellizzi V, Russo R, Chiodini P, Minutolo R, Conte G, De Nicola L. Incremental dialysis in ESRD: systematic review and meta-analysis. J Nephrol. 2019 Oct;32(5):823-836. doi: 10.1007/s40620-018-00577-9. Epub 2019 Jan 2. PMID 30604150
- [Background] Ronco C, Verger C, Crepaldi C, Pham J, De Los Rios T, Gauly A, Wabel P, Van Biesen W; IPOD-PD Study Group. Baseline hydration status in incident peritoneal dialysis patients: the initiative of patient outcomes in dialysis (IPOD-PD study)dagger. Nephrol Dial Transplant. 2015 May;30(5):849-58. doi: 10.1093/ndt/gfv013. Epub 2015 Mar 11. PMID 25762355
- [Background] Guo Q, Yi C, Li J, Wu X, Yang X, Yu X. Prevalence and risk factors of fluid overload in Southern Chinese continuous ambulatory peritoneal dialysis patients. PLoS One. 2013;8(1):e53294. doi: 10.1371/journal.pone.0053294. Epub 2013 Jan 14. PMID 23341936
- [Background] Guo Q, Lin J, Li J, Yi C, Mao H, Yang X, Yu X. The Effect of Fluid Overload on Clinical Outcome in Southern Chinese Patients Undergoing Continuous Ambulatory Peritoneal Dialysis. Perit Dial Int. 2015 Dec;35(7):691-702. doi: 10.3747/pdi.2014.00008. Epub 2015 Jul 7. PMID 26152580
- [Background] Agar BU, Sloand JA. Single Daily Icodextrin Exchange as Initial and Solitary Therapy. Perit Dial Int. 2018 Mar-Apr;38(2):119-124. doi: 10.3747/pdi.2017.00130. Epub 2018 Jan 31. PMID 29386305
- [Background] Goossen K, Becker M, Marshall MR, Buhn S, Breuing J, Firanek CA, Hess S, Nariai H, Sloand JA, Yao Q, Chang TI, Chen J, Paniagua R, Takatori Y, Wada J, Pieper D. Icodextrin Versus Glucose Solutions for the Once-Daily Long Dwell in Peritoneal Dialysis: An Enriched Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Kidney Dis. 2020 Jun;75(6):830-846. doi: 10.1053/j.ajkd.2019.10.004. Epub 2020 Feb 4. PMID 32033860
- [Background] Guest S, Leypoldt JK, Cassin M, Schreiber M. Kinetic Modeling of Incremental Ambulatory Peritoneal Dialysis Exchanges. Perit Dial Int. 2017 Mar-Apr;37(2):205-211. doi: 10.3747/pdi.2016.00055. Epub 2017 Jan 17. PMID 28096442
- [Background] Boateng EA, East L. The impact of dialysis modality on quality of life: a systematic review. J Ren Care. 2011 Dec;37(4):190-200. doi: 10.1111/j.1755-6686.2011.00244.x. PMID 22035363
- [Background] Davies SJ, Phillips L, Griffiths AM, Russell LH, Naish PF, Russell GI. What really happens to people on long-term peritoneal dialysis? Kidney Int. 1998 Dec;54(6):2207-17. doi: 10.1046/j.1523-1755.1998.00180.x. PMID 9853287